CLINICAL TRIAL: NCT03265067
Title: Field Implementation of the autoRIC Device in STEMI
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Osler Health System (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Trillium Health Centre (Other); Peel Regional Paramedic Service (Unknown); Halton Region Paramedic Services (Other); CellAegis US, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Sheldon Cheskes, Medical Director, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 16-0008
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Before and after phase study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Before' group (No Intervention): Patients who underwent primary PCI for STEMI prior to implementation of the RIC protol. These patients were not treated with the autoRIC device prior to PCI.
- 'After' group (Experimental): Patients who underwent primary PCI for STEMI after implementation of the RIC protocol. These patients were treated with the autoRIC device prior to PCI.
  Interventions: Device: autoRIC

INTERVENTIONS:
Device: autoRIC — Application of the autoRIC device
  Arms: 'After' group

SUMMARY:
This is a "before and after" observational study of a therapeutic strategy to treat patients with confirmed ST-segment myocardial infarction (STEMI) with remote ischemic conditioning (RIC) before undergoing primary percutaneous coronary intervention (PCI). RIC is the purposeful application of brief, intermittent cycles of limb occlusion by inflation/deflation of a pneumatic cuff. The autoRIC device is an automatic RIC delivery device (the autoRIC® Device; CellAegis Devices Inc, Toronto, ON) that has received clearance from Health Canada for this use under the direction of a health care professional. Paramedics in the Peel and Halton regional emergency services and the Emergency department (ED) staff of Brampton Civic Hospital and Mississauga Hospital will treat patients experiencing STEMI with autoRIC, and study data will be collected from existing patient records.

The 'before' group will include up to 900 patients who were treated before autoRIC implementation in the services and hospitals. These patients would have had a STEMI and undergone PCI, but did not receive the autoRIC device. The 'after' group will include up to 900 eligible patients who have had RIC treatment with the autoRIC device at the two participating sites following implementation in the services and hospitals.

The primary analyses will compare the short-term and long-term outcomes of eligible patients who have received completed primary PCI for STEMI in the time period before the implementation and following the implementation of this RIC strategy. In addition, a health economic analysis will be conducted to determine the cost-effectiveness of the therapeutic strategy to treat STEMI patients with RIC prior to PCI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older;
* patients diagnosed with STEMI in the prehospital environment by responding paramedics from Peel Regional Paramedic Services or Halton Emergency Medical Service and transported to the PCI laboratory of Brampton Civic Hospital or Trillium Health Partners;
* walk-in patients diagnosed with STEMI in the ED of either of these two facilities.

Exclusion Criteria:

* left-bundle branch block;
* Lymphedema on either arm
* PICC Line on either arm
* AV fistula or no palpable pulse on either arm;
* patient has a known bleeding disorder or known abnormality of blood flow to the left arm;
* patient has peripheral nerve injury, abnormal nerve supply, peripheral neuropathy or pre- existing traumatic injury to the limb to be treated (left-arm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1622 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
90-day MACCE | Within 90 days of PCI
  Major adverse cardiovascular and cerebrovascular events (MACCE) in-hospital and within 90 days of PCI.

SECONDARY OUTCOMES:
30, 60 and 180-day MACCE | Within 30, 60 and 180 days of admission
  MACCE within 30, 60 and 180 days post hospital admission
LOS | Time from hospital admission to hospital discharge, up to 180 days of admission
  Index hospitalization length of stay (LOS)
Cardiovascular-related death | Time from hospital admission to hospital discharge, up to 180 days of admission
  Death due to cardiovascular related events
30, 60, and 180-day cardiovascular-related readmission | 30, 60 and 180 days after index hospitalization
  Hospital readmission within 30, 60, and 180 days of index hospitalization, due to cardiovascular events.
Infarct size | Time from hospital admission to hospital discharge, up to 180 days of admission
  Size of infarct as measured by peak troponin level during index event admission

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Brampton Civic Hospital, Brampton, Ontario
  - The Mississauga Hospital, Mississauga, Ontario

IPD SHARING:
Plan to Share IPD: No